CLINICAL TRIAL: NCT01139086
Title: Role of Endothelial Function, Muscular Fitness and Metabolism in Functional Activity in Patients With Chronic Heart Failure
Brief Title: Role of Endothelial Function, Muscular Fitness and Metabolism in Functional Activity in Patients With Chronic Heart Failure (CHF)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ying-Tai Wu, School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University
Other Study IDs: 201003050R
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Heart Failure; Coronary Disease; Dilated Cardiomyopathy
Keywords: chronic heart failure; isokinetic test; near-infrared spectroscopy; laser Doppler flowmetry; endothelial function
MeSH Terms: conditions — Coronary Disease; Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cardiovascular disease: Diagnosis of cardiomyopathy or ischemic heart disease without heart failure
- Chronic heart failure: Diagnosis of cardiomyopathy or ischemic heart disease LVEF <40%
- Control: Age and body built matched with chronic heart failure group

SUMMARY:
Shortness of breath, fatigue, and exercise intolerance are clinical symptoms of chronic heart failure (CHF). Recent studies suggested that peripheral impairment was the major cause of clinical symptoms, and mechanism may be related to neuroendocrine impairment and vascular smooth muscle dysfunction. It results in increased peripheral resistance that may influence limb blood flow, muscle fitness and activities of daily.The purposes of this study are

1. to compare muscular strength, endurance, and perfusion of quadriceps between CHF patients and healthy controls by isokinetic test and near-infrared spectroscopy (NIRS) and difference in activities of daily living
2. to compare endothelium function between CHF patients and healthy control subjects
3. the relationship between endothelium function, muscular strength, endurance, perfusion, and metabolism of quadriceps.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75 years
* Chronic heart failure: ejection fraction<40% and at stable condition
* Coronary Disease and dilated cardiomyopathy without heart failure
* Control group without diagnosis of any heart disease

Exclusion Criteria:

* Clinical diagnosis of neuromusculoskeletal , pulmonary, or other systemic diseases that may affect the testing of the study

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic Heart Failure Coronary Disease Dilated Cardiomyopathy Control group without diagnosis of any heart disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
muscle strength and endurance | baseline
  Measured by biodex

SECONDARY OUTCOMES:
skeletal muscle oxygenation response | baseline
  Measured by near-infrared spectroscopy
Walking distance in 6-minute walking test | baseline
  walking distance (m)
laser Doppler flowmetry combine iontophoresis | baseline
  To measure the blood flux (PU) response to Ach (endothelial-dependent agent) and SNP (endothelial-independent agent)
sit-to-stand test | baseline
  Measured times in 1 minute
questionnaire (functional activity and quality of life) | baseline
Analysis of venous blood sample | baseline
  By standard venipuncture

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan